CLINICAL TRIAL: NCT02229968
Title: Efficacy of ε-Aminocaproic Acid (EACA) in Children Undergoing Craniofacial Reconstruction Surgery
Brief Title: Efficacy of Amicar for Children Having Craniofacial Surgery
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO00004263
Record Dates: First submitted 2014-08-28; First posted 2014-09-03 (Estimated); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Craniosynostosis
Keywords: craniosynostosis; craniofacial; amicar; epsilon aminocaproic acid; ε-aminocaproic acid
MeSH Terms: conditions — Craniosynostoses | interventions — Aminocaproic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amicar (ε-aminocaproic acid) (Experimental): Treatment group 1: Amicar 100 mg/kg (0.4 mL/kg) IV loading dose, followed by an intraoperative continuous infusion at 40 mg/kg/hr (0.16 mL/kg/hr) to be continued until skin closure.
  Interventions: Drug: Amicar (ε-aminocaproic acid)
- normal saline (Placebo Comparator): Treatment group 2: Equal volume of normal saline (placebo control) at the same rate as treatment group 1.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Amicar (ε-aminocaproic acid)
  Other Names: Amicar; 6-aminohexanoic acid; epsilon aminocaproic acid
  Arms: Amicar (ε-aminocaproic acid)
Drug: normal saline
  Other Names: normal saline 0.9%; placebo; placebo control
  Arms: normal saline

SUMMARY:
The purpose of this study is to determine whether Amicar (ε-aminocaproic acid) is effective in reducing blood loss in children undergoing craniofacial reconstruction surgery.

The investigators hypothesize that Amicar will decrease intraoperative blood loss and decrease the need for perioperative blood product administration in children undergoing craniofacial surgery.

DETAILED DESCRIPTION:
Craniosynostosis is a condition in which there is premature fusion of one or more of the sutures between the bones of the skull. Premature fusion of sutures in the skull limits the ability of the cranial vault to expand to accommodate the rapidly growing brain in infancy and early childhood and leads to bony deformation. Left uncorrected, craniosynostosis may adversely impact both neurologic and psychosocial development and in some cases, can result in high intracranial pressure and blindness.

Craniofacial (CF) reconstructive surgery is performed in young children with craniosynostosis to improve physical appearance, prevent functional neurologic disturbances, and enhance psychosocial development. Due to the complexities of the surgery as well as the young age and size of the patients, CF reconstruction carries potential life threatening risks and can result in significant morbidity. Reported complications include massive intraoperative hemorrhage, intraoperative cardiac arrest, transfusion-related reactions, venous air embolism, hypotension, coagulopathy, bradycardia, postoperative seizures, surgical site infections, facial swelling with airway compromise, and unplanned postoperative mechanical ventilation. The most severe and most common perioperative issues relate to the rate and extent of blood loss.

Fibrinolysis, which impairs adequate hemostasis, has been shown to occur in children during CF reconstruction. This most certainly contributes to the magnitude of blood loss in these types of operations. Thus, targeting this defect in clot hemostasis with the use of antifibrinolytics is a reasonable therapeutic approach.

Amicar (ε-aminocaproic acid) is a synthetic lysine analog that blocks the lysine binding sites on plasminogen, resulting in antifibrinolytic activity through inhibition of plasmin formation. We have chosen to study Amicar in this clinical context for a number of reasons. First, major hemorrhage continues to be a significant perioperative issue in this cohort. Secondly, Amicar is commonly and safely administered to children undergoing other types of high-risk surgery (i.e., spinal fusion surgery and open heart surgery). In addition, Amicar is inexpensive and easily administered, making it a viable and novel therapeutic option if shown to be effective for this type of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Any child diagnosed with craniosynostosis in need of surgical repair
* Males and females between the ages of 2 - 36 months (minorities will be included)
* Surgical procedure involving complex craniofacial reconstruction and craniotomy
* Written informed consent from parent/guardian

Exclusion Criteria:

* Subjects with known or suspected hypersensitivity reaction to Amicar or history of prior Amicar exposure
* Presence or prior history of a known coagulation disorder or hypercoagulable state
* Preoperative laboratory values that indicate clinically significant hematologic disease (hemoglobin, platelet count, prothrombin time, or partial thromboplastin time outside of normal range)
* Subjects who are on anticoagulant therapy (Coumadin, heparin, aspirin, etc.)
* Subjects with a prior history of a thrombotic event
* History of renal malformation
* Presence of hematuria
* History of abnormal renal function - serum creatinine or blood urea nitrogen (BUN) value greater than 1.5 times the upper limit of the normal range
* Craniofacial reconstruction surgery performed in conjunction with an additional surgical procedure associated with blood loss
* Subjects who have been previously enrolled in this protocol may not be enrolled again

Ages: 2 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2014-10; Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood loss | within the first 72 hours after surgery
  As estimated blood loss is known to be inaccurate in this setting, mean intraoperative blood loss (in mL/kg) will be calculated using a formula previously described in this population.

SECONDARY OUTCOMES:
Blood donor exposure | within the first 30 days after surgery
  To establish that intraoperative administration of Amicar decreases perioperative blood donor exposure and need for transfusion following craniofacial reconstructive surgery

CONTACTS AND LOCATIONS:
Overall Officials: Srijaya K Reddy, MD, MBA, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stricker PA, Zuppa AF, Fiadjoe JE, Maxwell LG, Sussman EM, Pruitt EY, Goebel TK, Gastonguay MR, Taylor JA, Bartlett SP, Schreiner MS. Population pharmacokinetics of epsilon-aminocaproic acid in infants undergoing craniofacial reconstruction surgery. Br J Anaesth. 2013 May;110(5):788-99. doi: 10.1093/bja/aes507. Epub 2013 Jan 25. PMID 23353035
- [Background] Faberowski LW, Black S, Mickle JP. Blood loss and transfusion practice in the perioperative management of craniosynostosis repair. J Neurosurg Anesthesiol. 1999 Jul;11(3):167-72. doi: 10.1097/00008506-199907000-00002. PMID 10414670
- [Background] Stricker PA, Shaw TL, Desouza DG, Hernandez SV, Bartlett SP, Friedman DF, Sesok-Pizzini DA, Jobes DR. Blood loss, replacement, and associated morbidity in infants and children undergoing craniofacial surgery. Paediatr Anaesth. 2010 Feb;20(2):150-9. doi: 10.1111/j.1460-9592.2009.03227.x. PMID 20078812
- [Background] Henry DA, Carless PA, Moxey AJ, O'Connell D, Stokes BJ, Fergusson DA, Ker K. Anti-fibrinolytic use for minimising perioperative allogeneic blood transfusion. Cochrane Database Syst Rev. 2011 Mar 16;2011(3):CD001886. doi: 10.1002/14651858.CD001886.pub4. PMID 21412876
- [Background] Oppenheimer AJ, Ranganathan K, Levi B, Strahle JM, Kapurch J, Muraszko KM, Buchman SR. Minimizing transfusions in primary cranial vault remodeling: the role of aminocaproic acid. J Craniofac Surg. 2014 Jan;25(1):82-6. doi: 10.1097/SCS.0b013e3182a2e23f. PMID 24240766